CLINICAL TRIAL: NCT05623410
Title: A Randomized, Double-Blind, Active-Control, Multicenter, Phase 3 Study to Evaluate the Efficacy and Safety of "ATGC-110" Compared to "Xeomin®" in Patients Who Need Moderate or Severe Glabellar Line Improvement
Brief Title: Study to Compare the Efficacy and Safety of ATGC-110 (Botulinum Toxin) With Xeomin® for the Treatment of Moderate to Severe Glabellar Frown Lines
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ATGC Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBAP-PLN-002
Record Dates: First submitted 2022-11-13; First posted 2022-11-21 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Glabellar Frown Lines
MeSH Terms: interventions — Botulinum Toxins, Type A; incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botulinum toxin type A(ATGC-110) (Experimental): ATGC-110 will be injected to 5 glabellar lines (Each 4U/0.1ml, Total 20U/0.5ml)
  Interventions: Biological: ATGC-110
- Incobotulinumtoxin A (Xeomin®) (Active Comparator): Xeomin® will be injected to 5 glabellar lines (Each 4U/0.1ml, Total 20U/0.5ml)
  Interventions: Biological: Xeomin®

INTERVENTIONS:
Biological: ATGC-110 — ATGC-110 is a prescription medicine that is injected into muscles and used to improve the moderate to severe glabellar lines. It should be reconstituted with sterile, preservative-free 0.9% saline before use.
  Other Names: Clostridium Botulinum Type A
  Arms: Botulinum toxin type A(ATGC-110)
Biological: Xeomin® — Xeomin® is a prescription medicine that is injected into muscles and used to improve the moderate to severe glabellar lines. It should be reconstituted with sterile, preservative-free 0.9% saline before use.
  Other Names: Incobotulinumtoxin A
  Arms: Incobotulinumtoxin A (Xeomin®)

SUMMARY:
Efficacy and safety of the investigational product, ATGC-110, was evaluated in comparison with Xeomin for a total of 16 weeks after the administration in treatment of glabellar frown lines.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged between 19 to 65 years
* Subjects assigned a glabellar line severity grade of 2 or greater (moderate) at maximum frown assessed by the Investigator
* Subjects who provide written consent to voluntarily participate in the study after receiving and understanding a detailed explanation of the study

Exclusion Criteria:

* Subjects with diseases that may affect neuromuscular function, such as Myasthenia gravis, Lambert-Eaton syndrome, Amyotrophic lateral sclerosis, or motor neuropathy etc.)
* Subjects with the history of eyelid paralysis or ptosis
* Subjects with significant facial asymmetry
* Subjects whose glabellar lines cannot be satisfactorily improved with physical methods since lines are not flattened even using hands
* Infection, dermatological condition or scar at the treatment injection sites
* Subjects currently suffering acute diseases
* Subjects with the history of excessive alcohol consumption or drug addiction
* Condition including anxiety disorder, or any other significant psychiatric disorder (e.g. depression), in the investigator's opinion
* Subjects with concomitant illnesses that make them unsuitable for participation in the study by the Investigator such as malignant tumors, immunodeficiency (immune deficiency), kidney disease, liver disease, or lung disease
* Subjects with the history of treatment of the glabellar region (including the forehead) such as face lifting, permanent implants, or fillers
* Subjects who have received other procedures that may affect the assessment of the glabellar or forehead lines during the following periods; Within 6 months of screening: main ingredient hyaluronic acid skin filler, dermal resurfacing, chemical/mechanical skin peeling, skin peeling, Dermal photorejuvenation; Within 12 months of screening: Dermal fillers other than the main ingredient hyaluronic acid, nonpermanent soft tissue fillers
* Subjects who have received medication that inhibits neuromuscular function within the 4 weeks prior to screening such as muscle relaxants, anticholinergics, benzodiazepines and similar drugs, benzamides, tetracycline antibiotics, lincomycin antibiotics, and aminoglycoside antibiotics
* Subjects who have taken retinoid drugs (Isotretinoin, Alitretinoin, etc.) during the following period; Oral and systemic use: within 6 months of screening Topical applied on the face: within 3 months of screening
* Subjects who have received aspirin or NSAIDs within 7 days prior to administration of the IP (Use of low-dose aspirin (325 mg/day or less) to prevent blood clotting is allowed).
* Subjects taking anticoagulants or antiplatelet agents (Use of low-dose aspirin (325 mg/day or less) to prevent blood clotting is allowed)
* Subjects who are allergic or sensitive to the IP or its components
* Subjects who have received botulinum toxin preparations within 6 months from the time of screening
* Female subjects of childbearing age who do not agree to practice contraception using medically allowed contraceptive methods during the study period (hormonal contraception, IUD (intrauterine device) or IUS (intrauterine system), tubal ligation, dual protection (using a combination of male condom, female condom, cervical cap, contraceptive diaphragm, or contraceptive sponge)
* Pregnant or lactating women
* Subjects planning a facial cosmetic procedure (skin fillers, photorejuvenation, chemical/mechanical peeling, etc.) during the study period
* Subjects who have participated in other clinical trials within 30 days prior to participating in this study and have received an IP or medical device during the previous clinical studies
* Subjects directly related to the investigator (e.g. a dermatologist or plastic surgeon)
* Individuals who are not eligible for this study for any reason as per the Investigator's discretion

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-02-10 (Estimated); Study Completion 2023-06-10 (Estimated)

PRIMARY OUTCOMES:
Improvement rate (%) of glabellar lines at maximum frown according to the investigator's on-site evaluation at week 4 compared to the baseline | 4 weeks after the administration
  Investigators will assess subjects' glabellar lines with Facial Wrinkle Scale (FWS) at maximal frown; 0=none, 1=mild, 2=moderate or 3=severe.
  Only the subjects whose FWS score is 0- or 1-grade when it's assessed and ≥ 2-grade improvement from baseline will be defined as their glabellar lines are improved.

SECONDARY OUTCOMES:
Improvement rate (%) of glabellar lines at maximum frown according to the investigator's on-site evaluation at weeks 8, 12, and 16 compared to the baseline | 8, 12 and 16 weeks after the administration
  Investigators will assess subjects' glabellar lines with Facial Wrinkle Scale (FWS) at maximal frown; 0=none, 1=mild, 2=moderate or 3=severe.
  Only the subjects whose FWS score is 0- or 1-grade when it's assessed and ≥ 2-grade improvement from baseline will be defined as their glabellar lines are improved.
Improvement rate (%) of glabellar lines at rest according to the investigator's on-site evaluation at weeks 4, 8, 12, and 16 compared to the baseline | 4, 8, 12 and 16 weeks after the administration
  Investigators will assess subjects' glabellar lines with Facial Wrinkle Scale (FWS) at rest; 0=none, 1=mild, 2=moderate or 3=severe.
  Only the subjects whose FWS score is 0- or 1-grade when it's assessed and ≥ 2-grade improvement from baseline will be defined as their glabellar lines are improved.
Improvement rate (%) of glabellar lines at maximum frown evaluated through photographs by the independent evaluator at weeks 4, 8, 12, and 16 compared to the baseline | 4, 8, 12 and 16 weeks after the administration
  Independent evaluator will assess subjects' glabellar lines with Facial Wrinkle Scale (FWS) at maximal frown; 0=none, 1=mild, 2=moderate or 3=severe.
  Only the subjects whose FWS score is 0- or 1-grade when it's assessed and ≥ 2-grade improvement from baseline will be defined as their glabellar lines are improved.
Improvement rate (%) of glabellar lines at rest evaluated through photographs by the independent evaluator at weeks 4, 8, 12, and 16 compared to the baseline | 4, 8, 12 and 16 weeks after the administration
  Independent evaluator will assess subjects' glabellar lines with Facial Wrinkle Scale (FWS) at rest; 0=none, 1=mild, 2=moderate or 3=severe.
  Only the subjects whose FWS score is 0- or 1-grade when it's assessed and ≥ 2-grade improvement from baseline will be defined as their glabellar lines are improved.
The percentage of subjects whose FWS score is 0- or 1-grade at maximal frown according to the investigator's on-site evaluation at week 4, 8, 12, and 16 | 4, 8, 12 and 16 weeks after the administration
  Investigators will assess subjects' glabellar lines with Facial Wrinkle Scale (FWS) at maximal frown; 0=none, 1=mild, 2=moderate or 3=severe.
The percentage of subjects whose FWS score is 0- or 1-grade at rest according to the investigator's on-site evaluation at week 4, 8, 12, and 16 | 4, 8, 12 and 16 weeks after the administration
  Investigators will assess subjects' glabellar lines with Facial Wrinkle Scale (FWS) at rest; 0=none, 1=mild, 2=moderate or 3=severe.
The percentage of subjects whose FWS score is 0- or 1-grade at maximal frown evaluated through photographs by the independent evaluator at week 4, 8, 12, and 16 | 4, 8, 12 and 16 weeks after the administration
  Independent evaluator will assess subjects' glabellar lines with Facial Wrinkle Scale (FWS) at rest; 0=none, 1=mild, 2=moderate or 3=severe.
The percentage of subjects whose FWS score is 0- or 1-grade at rest evaluated through photographs by the independent evaluator at week 4, 8, 12, and 16 | 4, 8, 12 and 16 weeks after the administration
  Independent evaluator will assess subjects' glabellar lines with Facial Wrinkle Scale (FWS) at rest; 0=none, 1=mild, 2=moderate or 3=severe.
The percentage of subjects whose FWS score is improved ≥ 2 grade improvement according to the subject's evaluation at week 4, 8, 12, and 16 | 4, 8, 12 and 16 weeks after the administration
  Subjects will assess their glabellar lines with Facial Wrinkle Scale (FWS) at rest; 0=none, 1=mild, 2=moderate or 3=severe.
Evaluation of subjects' satisfaction at weeks 4, 8, 12, and 16 | 4, 8, 12 and 16 weeks after the administration
  If the subject's satisfaction evaluation score is 6 points or higher, it is evaluated as satisfactory.
The percentage of subjects whose FWS score is imporved ≥ 2 grade improvement at maximal frown according to the investigator's on-site and subject's evaluation at weeks 4, 8, 12, and 16 | 4, 8, 12 and 16 weeks after the administration
  If the glabellar line score evaluated by the subject is +2 points or higher, it is evaluated as improved

CONTACTS AND LOCATIONS:
Locations (1):
- Nowon Eulji Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No